CLINICAL TRIAL: NCT07389291
Title: Effectiveness of Liuzijue and Box Breathing Techniques on Inspiratory Capacity and Blood Pressure Following Femoral Neck Fracture Immobilization: A Retrospective Comparative Study
Brief Title: Effect of Liuzijue and Box Breathing on Inspiratory Capacity and Blood Pressure After Femoral Neck Fracture Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Srivatsan Munusamy, Principal Investigator, Saveetha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 065/05/2025/ISRB/PGSR/SCPT
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Femoral Neck Fractures; Breathing Exercises; Inspiratory Capacity; Blood Pressure
Keywords: Femoral Neck Fractures; Qi Gong; Good Health and Well-Being; Aged
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liuzijue Qi Gong Exercise Group (Experimental)
  Interventions: Other: Liuzijue Qi Gong Exercise
- Box Breathing Technique Group (Active Comparator)
  Interventions: Other: Box Breathing Technique

INTERVENTIONS:
Other: Liuzijue Qi Gong Exercise — Liuzijue Qi Gong is a gentle breathing exercise from traditional Chinese medicine. It involves six specific vocal sounds ("Xu", "He", "Hu", "Si", "Chui", and "Xi"). The practice promotes deep, diaphragmatic breathing, improves lung function and supports relaxation. Participants performed Liuzijue Qi Gong exercises for 20 minutes, twice daily, 6 days per week, for 4 weeks following femoral neck fracture.
  Other Names: Six Character Qi Gong
  Arms: Liuzijue Qi Gong Exercise Group
Other: Box Breathing Technique — Box Breathing is a controlled breathing exercise that involves four equal phases: inhale, hold, exhale, hold, typically performed for 4-6 seconds each. It helps regulate breathing, reduce stress, improve oxygenation, and enhance autonomic balance. Safely practiced by older adults or individuals with limited physical activity. Participants performed the Box Breathing technique for 20 minutes, twice daily, 6 days per week, for 4 weeks following femoral neck fracture.
  Other Names: Four-Square Breathing
  Arms: Box Breathing Technique Group

SUMMARY:
The purpose of this study is to understand how two simple breathing exercise techniques (Liuzijue and box breathing) affect inspiratory capacity and blood pressure in people who were immobilized after a femoral neck fracture.

Older adults who sustain a femoral neck fracture are often required to remain immobile for several weeks. Prolonged immobilization can reduce lung capacity and may negatively affect blood pressure control, increasing the risk of breathing difficulties and other health problems. Breathing-based exercise techniques may help improve respiratory function and cardiovascular stability during recovery.

This study retrospectively analyzed data from patients who had previously received either Liuzijue exercises or box breathing techniques as part of their rehabilitation program. The main questions this study aimed to answer were:

Do Liuzijue and box breathing techniques improve inspiratory capacity after a period of immobilization? Do these techniques help in controlling systolic and diastolic blood pressure? Is one technique more effective than the other over a 4-week intervention period?

Data were collected at three time points: before the intervention (baseline), at the second week, and at the end of the fourth week. The findings of this study may help healthcare professionals choose simple, safe, and cost-effective breathing interventions for patients recovering from femoral neck fractures.

DETAILED DESCRIPTION:
Femoral neck fractures are common in the elderly population and are frequently associated with prolonged periods of immobilization. Extended immobilization can lead to reduced lung volumes, impaired inspiratory capacity and alterations in blood pressure regulation due to decreased physical activity and respiratory muscle disuse. These changes increase the risk of respiratory complications and cardiovascular instability during recovery.

Liuzijue is a traditional breathing-based exercise that combines slow, controlled breathing with specific vocalized exhalation patterns. It has been shown to improve respiratory muscle function, lung volumes and autonomic regulation. Box Breathing is a simple, structured breathing technique involving equal phases of inhalation, breath-holding, exhalation, and breath-holding and is known to promote relaxation and cardiovascular stability through autonomic nervous system modulation.

This retrospective study analyzed data from patients who had undergone a 4-week breathing-based intervention program following immobilization due to femoral neck fracture. Participants were divided into two groups based on the intervention they received: the Liuzijue exercise group and the Box Breathing technique group. Both interventions were administered for 20 minutes per session, twice daily, six days per week, over a period of four weeks as part of routine physiotherapy care.

Inspiratory capacity was measured using a volume-oriented incentive spirometer, while blood pressure parameters, including systolic and diastolic blood pressure, were recorded using a Digital sphygmomanometer. Outcome measures were documented at baseline (prior to intervention), at the end of the second week and at the completion of the fourth week.

The primary outcome of the study was the change in inspiratory capacity over the intervention period. Secondary outcomes included changes in systolic and diastolic blood pressure. Data were analyzed to evaluate within-group improvements over time and to compare the effectiveness of Liuzijue and Box Breathing techniques.

The findings of this study aim to provide evidence regarding the effectiveness of simple, non-invasive breathing-based interventions in improving respiratory function and blood pressure control in elderly individuals recovering from femoral neck fracture immobilization. The results may assist clinicians in selecting appropriate respiratory rehabilitation strategies for this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 65-85 years
* Femoral neck fracture managed conservatively or surgically.
* Volume-oriented incentive spirometer level less than 1000ml
* Blood pressure between 130/85 mmHg and 150/95 mmHg, not on regular antihypertensive medications
* Minimum 2 weeks of immobilization following the fracture.
* Ability to understand instructions and follow simple exercise routines.
* Ability to provide informed consent.

Exclusion Criteria:

* Recent major surgery (other than the femoral fracture)
* Severe hearing or speech impairment
* Uncontrolled hypertension (BP > 150/95 mmHg)
* Use of supplemental oxygen at rest
* Cognitive impairment
* History of cardiovascular events in the past 6 months
* History of recurrent syncope or dizziness
* Severe uncontrolled pain in the lower limb

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Inspiratory Capacity (mL) measured using Volume-Oriented Incentive Spirometer | Baseline (Pre-test), Week 2, Week 4
  Inspiratory capacity will be quantitatively measured in milliliters (mL) using a volume-oriented incentive spirometer. Participants will perform three maximal slow inspiratory efforts in an upright sitting position, and the highest recorded value will be used for analysis. Measurements will be collected using the same calibrated spirometer device for all participants to ensure consistency. Data will be recorded as continuous numerical values in milliliters and analyzed as within-group and between-group changes over time.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure (mmHg) measured using Digital Sphygmomanometer | Baseline (Pre-test), Week 2, Week 4
  Systolic blood pressure will be measured in millimeters of mercury (mmHg) using a calibrated digital sphygmomanometer. Measurements will be taken with the participant in a seated position after a minimum of five minutes of rest. Two readings will be recorded at each assessment point, and the average of the two readings will be used for analysis. Data will be analyzed as continuous numerical values to assess changes over time.
Change in Diastolic Blood Pressure (mmHg) measured using Digital Sphygmomanometer | Baseline (Pre-test), Week 2, Week 4
  Diastolic blood pressure will be measured in millimeters of mercury (mmHg) using a calibrated digital sphygmomanometer under standardized conditions. Two readings will be obtained at each time point, and the average value will be recorded for analysis. Measurements will be expressed as continuous variables and compared across assessment time points.

CONTACTS AND LOCATIONS:
Overall Officials: Shenbaga Sundaram Subramanian, Study Director — Saveetha college of physiotherapy, Saveetha Institute of Medical and Technical Sciences [SIMATS].
Locations (1):
- Saveetha Medical College and Hospital (SMCH), Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takac M. [Professor MUDr. Frantisek Por 70 years old]. Bratisl Lek Listy. 1969;51(5):521-2. No abstract available. Slovak. PMID 4893237
- [Background] Husberg C, Murphy P, Bjorgo E, Kalland KH, Kolsto AB. Cellular localisation and nuclear export of the human bZIP transcription factor TCF11. Biochim Biophys Acta. 2003 May 12;1640(2-3):143-51. doi: 10.1016/s0167-4889(03)00041-7. PMID 12729924
- [Background] Lopert R, Lang DL, Hill SR, Henry DA. Differential pricing of drugs: a role for cost-effectiveness analysis? Lancet. 2002 Jun 15;359(9323):2105-7. doi: 10.1016/S0140-6736(02)08911-0. PMID 12086780
- [Background] Maguire FW. Stevens-Johnson syndrome due to sulindac: a case report and review of the literature. Del Med J. 1981 Apr;53(4):193-7. No abstract available. PMID 7227578
- [Background] Xu S, Zhang D, He Q, Ma C, Ye S, Ge L, Zhang L, Liu W, Chen Z, Zhou L. Efficacy of Liuzijue Qigong in patients with chronic obstructive pulmonary disease: A systematic review and meta-analysis. Complement Ther Med. 2022 May;65:102809. doi: 10.1016/j.ctim.2022.102809. Epub 2022 Jan 29. PMID 35093513

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT07389291/Prot_SAP_000.pdf